CLINICAL TRIAL: NCT04267419
Title: Malondialdehyde and Nitrous Oxide as Salivary Biomarkers for Different Oral Lesions
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Maha Abdelkawy, Phd, principle investigator, Beni-Suef University
Other Study IDs: FDBSUREC/17022019/AM
Record Dates: First submitted 2020-02-09; First posted 2020-02-12 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Oral Lichen Planus; Oral Cancer; Leukoplakia; Oral Keratoses
Keywords: malondialdehyde; nitric oxide; salivary biomarkers
MeSH Terms: conditions — Lichen Planus, Oral; Mouth Neoplasms; Leukoplakia; Leukoplakia, Oral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- healthy Control: MDA and NO in saliva
  Interventions: Diagnostic Test: salivary biomarker
- keratosis: MDA and NO in saliva
  Interventions: Diagnostic Test: salivary biomarker
- leukoplakia: MDA and NO in saliva
  Interventions: Diagnostic Test: salivary biomarker
- Oral lichen Planus: MDA and NO in saliva
  Interventions: Diagnostic Test: salivary biomarker
- oral Squamous cell carcinoma: MDA and NO in saliva
  Interventions: Diagnostic Test: salivary biomarker

INTERVENTIONS:
Diagnostic Test: salivary biomarker — MDA and NO as salivary biomarkers

SUMMARY:
investigating the level of malondialdehyde (MDA) & nitric oxide (NO) in saliva in oral premalignant and malignant lesions in order to determine their diagnostic value for the malignant and potentially malignant lesions.

DETAILED DESCRIPTION:
Being a detrimental disease, cancer development is a very complicated process that requires many sequential steps and depends on a various number of genetic alterations and factors(1). Among these factors are the free radicals which are derived either from endogenous or exogenous sources (5). Free radicals result in an oxidative stress of the affected cells generating a body imbalance between oxidants and antioxidants (6).

In this regard, saliva has been currently used to assess this possible oxidative imbalance through various salivary biomarkers including nitric oxide (NO) and malondialdehyde (MDA). Saliva could be used as a very interesting rich medium, known for its role in diagnosis, prognosis and treatment that has become more prominent in oral diseases (6).

Nitric oxide (NO) is an intercellular messenger molecule having many important biological functions. The levels of nitric oxide in salivary secretions could be used to monitor the severity of many underlying disease processes. Moreover, malondialdehyde (MDA) has been the most frequently used biomarker of oxidative stress in many pathological conditions such as cancer. It resulted from reactive oxygen species lipid degradation and induced toxic stress in affected cells, making both biomarkers a point of focus in monitoring clinical progress of suspected lesions

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals with one of the following oral lesions :

  * keratosis
  * Oral lichen planus
  * oral squamous cell carcinoma
  * oral leukoplakia

Exclusion Criteria:

* subjects having systemic disorders
* pregnant or lactating females;
* subjects who suffered from any other mucosal lesions;
* severe periodontal inflammation.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: out patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Salivary MDA level in different oral lesions | 9 months
  The MDA level in saliva measured using ELISA kit provided by My BioSource, USA.
Salivary NO level in different oral lesions | 9 MONTHS
  The nitric oxide level in saliva measured using ELISA kit provided by My BioSource, USA.

CONTACTS AND LOCATIONS:
Overall Officials: weam Elbattawy, Phd, Principal Investigator — Cairo University
Locations (1):
- Maha Abdelkawy, Phd, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all the data will shared once the work is published
Supporting Information: Study Protocol, CSR
Time Frame: once published